CLINICAL TRIAL: NCT03856632
Title: Novel Medical Adjunctive Therapy to Catheter Ablation For Atrial Fibrillation (AF)
Brief Title: Liraglutide Effect in Atrial Fibrillation
Acronym: LEAF
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Jeffrey Goldberger, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20181182
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Liraglutide; Anti-Arrhythmia Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Risk Factor Modification (RFM) (Active Comparator): A structured risk factor modification (RFM) program currently offered to all patients who are overweight or obese undergoing an ablation procedure for atrial fibrillation.The RFM program is already offered through our Center for Atrial Fibrillation and is managed by a nurse practitioner. The RFM program will provide patient teaching and education on weight, fitness,blood pressure control, glucose control, cholesterol, sleep apnea, smoking, and alcohol.
  Interventions: Other: RFM; Drug: Anti Arrhythmics; Procedure: Afib Catheter Ablation
- RFM plus Liraglutide (Experimental): In addition to RFM, Liraglutide will be administered. Liraglutide is an FDA approved medication used as an adjunct to a reduced-calorie diet and increased physical activity for chronic weight management of obese adults with weight-related comorbid conditions.
  Interventions: Drug: Liraglutide; Other: RFM; Drug: Anti Arrhythmics; Procedure: Afib Catheter Ablation

INTERVENTIONS:
Drug: Liraglutide — Liraglutide will be administered with a starting dose of 0.6 mg once daily and subsequent increments to 1.2 mg once daily (after at least one week) and to 1.8 mg once daily (after at least a week on 1.2 mg). This will be taken for 3 consecutive months in conjunction with RFM program prior to catheter ablation. Treatment will resume post ablation and will be continue for 6 months.
  Arms: RFM plus Liraglutide
Other: RFM — The program involves weight management and exercise regimen (30 minutes for 2 to 4 times a week), hyperlipidemia management (lifestyle measure changes and initiation of statins and fibrates if necessary), management of obstructive sleep apnea (initiation of Continuous Positive Airway Pressure (CPAP) if necessary), management of hypertension (reduction of salt intake, initiation of Angiotensin Converting Enzyme Inhibitor (ACEI) or Angiotensin II Receptor blockers (ARB) medications if necessary), diabetes management (lifestyle measure changes, endocrine review and initiation of metformin if necessary) and smoking cessation and alcohol abstinence or reduction. This program will be performed at start of study participation all throughout the follow up period.
Drug: Anti Arrhythmics — The choice of antiarrhythmic drug will be at the discretion of the managing physician, but will generally include either a class IC or class III antiarrhythmic drug. If necessary, and clinically indicated, amiodarone may be used. Therapy will be initiated at the start of study participation and will be discontinued 6-12 weeks after the ablation, as deemed clinically appropriate by the managing electrophysiologist.
Procedure: Afib Catheter Ablation — The procedure will be performed according to usual clinical practice. The primary approach will be antral pulmonary vein isolation (PVI), preferably performed by cryoballoon ablation, though radiofrequency may be used as deemed necessary by the operator for clinical reasons. This will be performed after 3 months of RFM or RFM + Liraglutide program.

SUMMARY:
The goal (or purpose) of this study is to evaluate (study) a new way to stabilize (steady) the activity between the fat deposits surrounding the heart and the left atrium.

To reduce the amount of EAT, this study will use a medication called Liraglutide. This medication is known to work on fat deposits and produce weight loss. The investigator is conducting this study to find out if Liraglutide will reduce the fat deposits surrounding the participant's heart, and stabilize (and perhaps reduce or eliminate) atrial fibrillation activity.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, age 18 or older
* Persistent AF defined as continuous AF sustained beyond 7 days (or AF with the decision to cardiovert before 7 days of enrollment or Paroxysmal AF defined as recurrent AF (≥2 episodes) that terminates spontaneously within 7 days
* BMI ≥27 kg/m2
* Patient wishes to undergo a catheter ablation procedure for the treatment of atrial fibrillation
* Receiving follow-up care at the University of Miami

Exclusion Criteria:

* Inability to sign an informed consent
* Patients with longstanding persistent atrial fibrillation of more than 3 years
* Prior ablation for atrial fibrillation
* Patients not appropriate candidates for catheter ablation such as those with AF due to acute or chronic precipitating medical conditions, for example, hypothyroidism and hyperthyroidism, significant pulmonary disease, pulmonary embolism, left atrial thrombus, class IV heart failure)
* Patients with a life expectancy <1 year
* Patients with a serious medical condition (for example, recent cancer with chemotherapy or radiation therapy within 4 weeks before entering the study) who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Known contraindications to Liraglutide, such as the previous history of pancreatitis or medullary thyroid carcinoma
* Personal or family history of multiple endocrine neoplasias
* Known serious hypersensitivity reaction to Liraglutide
* Patients using, glitazones, sodium-glucose transporters 2 inhibitors (SGLT2i), other GLP-1 analogs, or DPP4 inhibitors
* Type 1 diabetes, defined by American Diabetes Association criteria, history of diabetic ketoacidosis, pancreas or beta-cell transplantation, or diabetes due to pancreatitis or pancreatectomy
* Poorly controlled type 2 diabetes with HbA1c > 10%
* Pregnant women
* Women who are breast-feeding or intend to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in size of Left Atrial Epicardial Adipose Tissue (LAEAT) | Baseline, 3 months (prior to ablation)
  As assessed via multi detector cardiac computer tomography (MD-CT)

SECONDARY OUTCOMES:
Change in size of Epicardial Adipose Tissue (EAT) thickness | Baseline, 3 months (prior to ablation), 1 year post-ablation
  As assessed via echocardiography
Change in atrial function | Baseline, 1 year post ablation
  As assessed via echocardiography
Change in atrial size | Baseline, 1 year post ablation
  As assessed via echocardiography
Change in C-Reactive Protein (CRP) value | Baseline, 1 year post ablation
  Serial changes in biomarkers of inflammation
Change in Interleukin-6 (IL-6) | Baseline, 1 year post ablation
  Serial changes in biomarkers of inflammation
Correlation of CRP expression in blood from left atrium to peripheral plasma | During the catheter ablation procedure
  At the same time point, blood will be collected directly from left atrium and peripheral vessel during the ablation procedure and compared
Correlation of IL-6 expression in blood from left atrium to peripheral plasma | During the catheter ablation procedure
  At the same time point blood, will be collected directly from left atrium and the peripheral vessel during the ablation procedure and compared
Correlation of plasminogen activator inhibitor (PAI-1), matrix metalloproteinase-2 (MMP2), Tissue inhibitor of metalloproteinase 2 (TIMP-2) | During the catheter ablation procedure
  At the same time point, blood will be collected directly from left atrium and the peripheral vessel during the ablation procedure and compared
Correlation of atrial natriuretic peptide (ANP), brain natriuretic peptide (BNP) | During the catheter ablation procedure
  At the same time point, blood will be collected directly from left atrium and the peripheral vessel during the ablation procedure and compared

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Goldberger, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No